CLINICAL TRIAL: NCT02835625
Title: Digital Breast Tomosynthesis - The Future Screening Tool for Breast Cancer?
Brief Title: The Digital Breast Tomosynthesis Trial in Bergen
Acronym: TOBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: Haukeland University Hospital (Other); University of Oslo (Other); The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 247941/H10
Record Dates: First submitted 2016-06-23; First posted 2016-07-18 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2020-01

CONDITIONS: Breast Neoplasms
Keywords: Diagnostic Imaging; Mammography; Randomized Controlled Trial; Tomosynthesis; Early performance measures; Recall; Radiation dose; Cancer detection; Sensitivity; Specificity; Cost; Economy
MeSH Terms: conditions — Breast Neoplasms; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Digital Breast Tomosynthesis (Active Comparator): Synthetic Mammography (SM) + Digital Breast Tomosynthesis (DBT)
  The SM+DBT will be independently read by two radiologists. A consensus meeting will decide whether to recall the woman or not.
  Women selected for further assessment (positive screening exam) will be recalled.
  Interventions: Radiation: Synthetic Mammography + Digital Breast Tomosynthesis
- Digital mammography (Active Comparator): The digital mammograms will be independently read by two radiologists. A consensus meeting will decide whether to recall the woman or not.
  Interventions: Radiation: Digital mammography

INTERVENTIONS:
Radiation: Synthetic Mammography + Digital Breast Tomosynthesis — Two-view tomosynthesis performed with GE Senoclaire 3D Breast Tomosynthesis.
  Other Names: SM+DBT
  Arms: Digital Breast Tomosynthesis
Radiation: Digital mammography — Two-view digital mammography performed with GE Senoclaire 3D Breast Tomosynthesis.
  Other Names: DM
  Arms: Digital mammography

SUMMARY:
Compare synthetic mammography+digital breast tomosynthesis (SM+DBT) with digital mammography (DM) as a screening tool for women aged 50-69 years, invited to participate in the Norwegian Breast Cancer Screening Program at the screening unit in Bergen, Norway, with regard to early performance measures, including prognostic and predictive tumor characteristics, radiation doses and cost-effectiveness.

DETAILED DESCRIPTION:
DBT is a new screening tool, argued to be better than standard DM. This statement is based on a lower recall rate, and a higher rate of early-stage screen-detected cancer. No studies have so far reported results from women screened with DBT from GE Healthcare, as far as the investigators know. DBT from GE offer synthetic two-dimensional DM generated from the DBT data (SM), and studies have shown similar detection rates for this technique as of adjacent DM. By comparing results of early performance measures and economic aspects in two comparable populations of women in the same age group, residing in the same county, the investigators can measure the effect of SM+DBT versus standard DM with equipment from GE Healthcare. The populations will be examined by the same radiographers, screen-read by the same radiologists, histologically breast cancer proven by the same pathologists, and treated by the same surgeons and oncologists.

A prospective cohort study targeting 45,000 women invited to breast cancer screening in Bergen, Hordaland in the study period, 2016-2018, will be performed. A screening participation of approximately 75% is expected. All attending women will be asked if they are willing to participate in the study after receiving written and oral information about the study. Women willing to participate in the study will sign an informed consent. Of the attending women it is expected that about 90-95% will consent to participate in the study. The women will be randomized into two groups, a study group and a control group. The randomization will take place at the screening unit in Bergen. The outcome of the randomization is based on the 11-digit personal identification number assigned to every citizen in Norway. In the study group, the women will be screened with SM+DBT. In the control group, the women will be screened with DM. Women not willing to participate in the study will be screened with DM, and not included in our study.

The investigators aim to address the following topics and research questions:

* Study 1: Early performance measures in a population based screening program using SM+DBT versus DM - interim analyses.
* Study 2: Use of SM+DBT versus DM in a population based screening program - a randomized controlled trial.
* Study 3: Prognostic and predictive histopathologic characteristics of breast tumors detected in a population based program using SM+DBT versus DM.
* Study 4: SM+DBT and DM in a populations based screening program - which technology has the highest sensitivity for women with mammographic dense breast?
* Study 5 and 6: Costs of SM+DBT and DM in a populations based screening program - is SM+DBT cost-effective?

ELIGIBILITY:
Inclusion Criteria:

* Informed consent

Exclusion Criteria:

* Breast implants

Ages: 48 Years to 71 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29453 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solveig Hofvind, Professor, Principal Investigator — Norwegian Institute of Public Health
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen, Hordaland
  - Cancer Registry of Norway, Oslo

IPD SHARING:
Plan to Share IPD: No
We will not share the data outside the project group

REFERENCES:
- [Background] Skaane P, Bandos AI, Gullien R, Eben EB, Ekseth U, Haakenaasen U, Izadi M, Jebsen IN, Jahr G, Krager M, Niklason LT, Hofvind S, Gur D. Comparison of digital mammography alone and digital mammography plus tomosynthesis in a population-based screening program. Radiology. 2013 Apr;267(1):47-56. doi: 10.1148/radiol.12121373. Epub 2013 Jan 7. PMID 23297332
- [Background] Ciatto S, Houssami N, Bernardi D, Caumo F, Pellegrini M, Brunelli S, Tuttobene P, Bricolo P, Fanto C, Valentini M, Montemezzi S, Macaskill P. Integration of 3D digital mammography with tomosynthesis for population breast-cancer screening (STORM): a prospective comparison study. Lancet Oncol. 2013 Jun;14(7):583-9. doi: 10.1016/S1470-2045(13)70134-7. Epub 2013 Apr 25. PMID 23623721
- [Background] Lang K, Andersson I, Rosso A, Tingberg A, Timberg P, Zackrisson S. Performance of one-view breast tomosynthesis as a stand-alone breast cancer screening modality: results from the Malmo Breast Tomosynthesis Screening Trial, a population-based study. Eur Radiol. 2016 Jan;26(1):184-90. doi: 10.1007/s00330-015-3803-3. Epub 2015 May 1. PMID 25929946
- [Background] Haas BM, Kalra V, Geisel J, Raghu M, Durand M, Philpotts LE. Comparison of tomosynthesis plus digital mammography and digital mammography alone for breast cancer screening. Radiology. 2013 Dec;269(3):694-700. doi: 10.1148/radiol.13130307. Epub 2013 Oct 28. PMID 23901124
- [Background] Durand MA, Haas BM, Yao X, Geisel JL, Raghu M, Hooley RJ, Horvath LJ, Philpotts LE. Early clinical experience with digital breast tomosynthesis for screening mammography. Radiology. 2015 Jan;274(1):85-92. doi: 10.1148/radiol.14131319. Epub 2014 Sep 1. PMID 25188431
- [Background] Friedewald SM, Rafferty EA, Rose SL, Durand MA, Plecha DM, Greenberg JS, Hayes MK, Copit DS, Carlson KL, Cink TM, Barke LD, Greer LN, Miller DP, Conant EF. Breast cancer screening using tomosynthesis in combination with digital mammography. JAMA. 2014 Jun 25;311(24):2499-507. doi: 10.1001/jama.2014.6095. PMID 25058084
- [Background] Rose SL, Tidwell AL, Bujnoch LJ, Kushwaha AC, Nordmann AS, Sexton R Jr. Implementation of breast tomosynthesis in a routine screening practice: an observational study. AJR Am J Roentgenol. 2013 Jun;200(6):1401-8. doi: 10.2214/AJR.12.9672. PMID 23701081
- [Background] McCarthy AM, Kontos D, Synnestvedt M, Tan KS, Heitjan DF, Schnall M, Conant EF. Screening outcomes following implementation of digital breast tomosynthesis in a general-population screening program. J Natl Cancer Inst. 2014 Oct 13;106(11):dju316. doi: 10.1093/jnci/dju316. Print 2014 Nov. PMID 25313245
- [Background] Greenberg JS, Javitt MC, Katzen J, Michael S, Holland AE. Clinical performance metrics of 3D digital breast tomosynthesis compared with 2D digital mammography for breast cancer screening in community practice. AJR Am J Roentgenol. 2014 Sep;203(3):687-93. doi: 10.2214/AJR.14.12642. Epub 2014 Jun 11. PMID 24918774
- [Background] Lourenco AP, Barry-Brooks M, Baird GL, Tuttle A, Mainiero MB. Changes in recall type and patient treatment following implementation of screening digital breast tomosynthesis. Radiology. 2015 Feb;274(2):337-42. doi: 10.1148/radiol.14140317. Epub 2014 Sep 22. PMID 25247407
- [Background] Destounis S, Arieno A, Morgan R. Initial experience with combination digital breast tomosynthesis plus full field digital mammography or full field digital mammography alone in the screening environment. J Clin Imaging Sci. 2014 Feb 25;4:9. doi: 10.4103/2156-7514.127838. eCollection 2014. PMID 24744966
- [Background] Skaane P, Bandos AI, Eben EB, Jebsen IN, Krager M, Haakenaasen U, Ekseth U, Izadi M, Hofvind S, Gullien R. Two-view digital breast tomosynthesis screening with synthetically reconstructed projection images: comparison with digital breast tomosynthesis with full-field digital mammographic images. Radiology. 2014 Jun;271(3):655-63. doi: 10.1148/radiol.13131391. Epub 2014 Jan 24. PMID 24484063
- [Background] Zuley ML, Guo B, Catullo VJ, Chough DM, Kelly AE, Lu AH, Rathfon GY, Lee Spangler M, Sumkin JH, Wallace LP, Bandos AI. Comparison of two-dimensional synthesized mammograms versus original digital mammograms alone and in combination with tomosynthesis images. Radiology. 2014 Jun;271(3):664-71. doi: 10.1148/radiol.13131530. Epub 2014 Jan 21. PMID 24475859
- [Background] Gilbert FJ, Tucker L, Gillan MG, Willsher P, Cooke J, Duncan KA, Michell MJ, Dobson HM, Lim YY, Suaris T, Astley SM, Morrish O, Young KC, Duffy SW. Accuracy of Digital Breast Tomosynthesis for Depicting Breast Cancer Subgroups in a UK Retrospective Reading Study (TOMMY Trial). Radiology. 2015 Dec;277(3):697-706. doi: 10.1148/radiol.2015142566. Epub 2015 Jul 15. PMID 26176654
- [Background] Houssami N, Skaane P. Overview of the evidence on digital breast tomosynthesis in breast cancer detection. Breast. 2013 Apr;22(2):101-108. doi: 10.1016/j.breast.2013.01.017. Epub 2013 Feb 16. PMID 23422255
- [Background] Bonafede MM, Kalra VB, Miller JD, Fajardo LL. Value analysis of digital breast tomosynthesis for breast cancer screening in a commercially-insured US population. Clinicoecon Outcomes Res. 2015 Jan 12;7:53-63. doi: 10.2147/CEOR.S76167. eCollection 2015. PMID 25624767
- [Background] Lee CI, Cevik M, Alagoz O, Sprague BL, Tosteson AN, Miglioretti DL, Kerlikowske K, Stout NK, Jarvik JG, Ramsey SD, Lehman CD. Comparative effectiveness of combined digital mammography and tomosynthesis screening for women with dense breasts. Radiology. 2015 Mar;274(3):772-80. doi: 10.1148/radiol.14141237. Epub 2014 Oct 28. PMID 25350548
- [Background] Moger TA, Bjornelv GM, Aas E. Expected 10-year treatment cost of breast cancer detected within and outside a public screening program in Norway. Eur J Health Econ. 2016 Jul;17(6):745-54. doi: 10.1007/s10198-015-0719-4. Epub 2015 Aug 4. PMID 26239280
- [Background] Tingberg A, Zackrisson S. Digital mammography and tomosynthesis for breast cancer diagnosis. Expert Opin Med Diagn. 2011 Nov;5(6):517-26. doi: 10.1517/17530059.2011.616492. Epub 2011 Sep 6. PMID 23484749
- [Result] Aase HS, Holen AS, Pedersen K, Houssami N, Haldorsen IS, Sebuodegard S, Hanestad B, Hofvind S. A randomized controlled trial of digital breast tomosynthesis versus digital mammography in population-based screening in Bergen: interim analysis of performance indicators from the To-Be trial. Eur Radiol. 2019 Mar;29(3):1175-1186. doi: 10.1007/s00330-018-5690-x. Epub 2018 Aug 29. PMID 30159620
- [Result] Hofvind S, Holen AS, Aase HS, Houssami N, Sebuodegard S, Moger TA, Haldorsen IS, Akslen LA. Two-view digital breast tomosynthesis versus digital mammography in a population-based breast cancer screening programme (To-Be): a randomised, controlled trial. Lancet Oncol. 2019 Jun;20(6):795-805. doi: 10.1016/S1470-2045(19)30161-5. Epub 2019 May 8. PMID 31078459
- [Result] Moger TA, Swanson JO, Holen AS, Hanestad B, Hofvind S. Cost differences between digital tomosynthesis and standard digital mammography in a breast cancer screening programme: results from the To-Be trial in Norway. Eur J Health Econ. 2019 Nov;20(8):1261-1269. doi: 10.1007/s10198-019-01094-7. Epub 2019 Aug 9. PMID 31399773
- [Result] Waade GG, Holen A, Sebuodegard S, Aase H, Pedersen K, Hanestad B, Hofvind S. Breast compression parameters among women screened with standard digital mammography and digital breast tomosynthesis in a randomized controlled trial. Acta Radiol. 2020 Mar;61(3):321-330. doi: 10.1177/0284185119863989. Epub 2019 Jul 25. No abstract available. PMID 31342757
- [Result] Moshina N, Aase HS, Danielsen AS, Haldorsen IS, Lee CI, Zackrisson S, Hofvind S. Comparing Screening Outcomes for Digital Breast Tomosynthesis and Digital Mammography by Automated Breast Density in a Randomized Controlled Trial: Results from the To-Be Trial. Radiology. 2020 Dec;297(3):522-531. doi: 10.1148/radiol.2020201150. Epub 2020 Sep 15. PMID 32930649
- [Result] Aase HS, Danielsen AS, Hoff SR, Holen AS, Haldorsen IS, Hovda T, Hanestad B, Sandvik CK, Hofvind S. Mammographic features and screening outcome in a randomized controlled trial comparing digital breast tomosynthesis and digital mammography. Eur J Radiol. 2021 Aug;141:109753. doi: 10.1016/j.ejrad.2021.109753. Epub 2021 May 5. PMID 34053786
- [Result] Hofvind S, Moshina N, Holen AS, Danielsen AS, Lee CI, Houssami N, Aase HS, Akslen LA, Haldorsen IS. Interval and Subsequent Round Breast Cancer in a Randomized Controlled Trial Comparing Digital Breast Tomosynthesis and Digital Mammography Screening. Radiology. 2021 Jul;300(1):66-76. doi: 10.1148/radiol.2021203936. Epub 2021 May 11. PMID 33973840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were invited to participate when attending screening at the screening unit Danmarksplass in Bergen, Norway. The recruitment period lasted from January 14th 2016 to December 15th 2017.
Pre-assignment Details: Women that attended screening but had breast implant were not invited to participate, and thus not randomized to either of the study groups.
Groups:
- Digital Breast Tomosynthesis: Digital Breast Tomosynthesis + Synthetic Mammography (DBT)
  The DBT was independently read by two radiologists. A consensus meeting decided whether to recall the woman or not.
  Women selected for further assessment (positive screening exam) was recalled.
  Digital Breast Tomosynthesis + Synthetic Mammography: Two-view tomosynthesis performed with GE SenoClaire 3D Breast Tomosynthesis.
- Digital Mammography: The digital mammograms was independently read by two radiologists. A consensus meeting decided whether to recall the woman or not.
  Women selected for further assessment (positive screening exam) was recalled.
  Digital mammography: Two-view digital mammography performed with GE SenoClaire 3D Breast Tomosynthesis.
Period: Overall Study
Arm/Group | Digital Breast Tomosynthesis | Digital Mammography
Started | 14734 | 14719
Completed | 14734 | 14719
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We excluded women with previous breast cancer (DBT = 314, DM = 316), women with breast symptoms at screening (DBT = 39, DM = 34) and one woman with metastasis from melanoma (DBT).
Groups:
- Total: Total of all reporting groups
Arm/Group | Digital Breast Tomosynthesis | Digital Mammography | Total
Number analyzed (Participants) | 14380 | 14369 | 28749
Age, Customized [Count of Participants; unit: Participants]
  <55 years | 3746 | 3813 | 7559
  55-59 years | 3628 | 3668 | 7296
  60-64 years | 3625 | 3492 | 7117
  >64 years | 3381 | 3396 | 6777
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14380 | 14369 | 28749
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Norway | 14380 | 14369 | 28749
Screening history [Count of Participants; unit: Participants]
  Prevalent (first screening) | 2013 | 2053 | 4066
  Subsequent | 12367 | 12316 | 24683

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Screen-Detected Breast Cancer
Description: Comparison of rates of screen-detected breast cancer in tomosynthesis versus digital mammography as performed in a population based screening program.
Time Frame: 36 months from start up of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Breast Tomosynthesis | Digital Mammography
Number analyzed (Participants) | 14380 | 14369
Participants | 95 | 87

2. Secondary Outcome: Number and Percentage of Participants Screen-Detected Breast Cancer Among Participants Recalled for Further Assesment
Description: Positive predictive value of recalls (number of screen-detected breast cancer among participants recalled for further assesment) for tomosynthesis versus digital mammography in a population based screening program.
Time Frame: 36 months from start up of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Breast Tomosynthesis | Digital Mammography
Number analyzed (Participants) | 444 | 571
Participants | 95 | 87

3. Secondary Outcome: Number of Participants Recalled for Further Assesment Due to Mammographic Findings
Description: Comparison of rate of recall for further assesment due to mammographic findings in tomosynthesis versus digital mammography as performed in a population based screening program.
Time Frame: 36 months from start up of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Breast Tomosynthesis | Digital Mammography
Number analyzed (Participants) | 14380 | 14369
Participants | 444 | 571

4. Secondary Outcome: Incremental Costs of Screening With Tomosynthesis Versus Digital Mammography
Description: The incremental cost per woman screened with digital breast tomosynthesis versus digital mammography in a population-based breast cancer screening program.
Time Frame: 36 months from start up of the trial
Population: For each participant, the incremental cost of tomosynthesis vs. digital mammography were estimated, not the total cost of tomosynthesis vs. digital mammography. The investigators assumed that costs not pertaining to examination and reading times, mammograph price, IT storage and connectivity were equal for the two. This Outcome Measure was pre-specified to present the incremental costs per screened woman. By nature, incremental costs are calculated between groups.
Measure: Mean (95% Confidence Interval); unit: €
Groups:
- Digital Breast Tomosynthesis Versus Digital Mammography: Comparing costs of procedure use and screening, recall and treatment costs estimated at the individual level for Digital Breast Tomosynthesis + Synthetic Mammography (DBT) versus Digital Mammography (DM).
Arm/Group | Digital Breast Tomosynthesis Versus Digital Mammography
Number analyzed (Participants) | 29453
€
  Incremental costs of DBT vs. DM in Euro | 8.5 [8.4 to 8.6]
  Incremental cost of DBT vs. DM after adding costs of recall, in Euro | 6.2 [4.6 to 7.9]

5. Secondary Outcome: Prognostic and Predictive Tumor Characteristics for Screen-Detected Breast Cancer
Description: Distribution of characteristics among the women diagnosed with breast cancer screened with tomosynthesis versus digital mammography in a population based screening program.
Time Frame: 36 months from start up of the trial
Population: When collecting information on histopathological tumor characteristics, not all participants had information available on all variables.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Breast Tomosynthesis | Digital Mammography
Number analyzed (Participants) | 80 | 71
Participants
  Histological type : Carcinoma (no special type) | 62 | 51
  Histological type : Lobular carcinoma | 6 | 13
  Histological type : Tubular carcinoma | 2 | 4
  Histological type : Other carcinoma | 10 | 3
  Tumor diameter : <10 mm: number analyzed (Participants) | 70 | 60
  Tumor diameter : <10 mm | 10 | 18
  Tumor diameter : >=10-<20 mm: number analyzed (Participants) | 70 | 60
  Tumor diameter : >=10-<20 mm | 43 | 29
  Tumor diameter : >=20 mm: number analyzed (Participants) | 70 | 60
  Tumor diameter : >=20 mm | 17 | 13
  Lymph node positive: number analyzed (Participants) | 79 | 70
  Lymph node positive | 14 | 18
  Histological grade : grade 1: number analyzed (Participants) | 76 | 69
  Histological grade : grade 1 | 22 | 24
  Histological grade : grade 2: number analyzed (Participants) | 76 | 69
  Histological grade : grade 2 | 38 | 35
  Histological grade : grade 3: number analyzed (Participants) | 76 | 69
  Histological grade : grade 3 | 16 | 10
  Estrogen receptor positive: number analyzed (Participants) | 79 | 71
  Estrogen receptor positive | 71 | 69
  Progesterone receptor positive: number analyzed (Participants) | 79 | 71
  Progesterone receptor positive | 61 | 62
  HER2 positive: number analyzed (Participants) | 79 | 71
  HER2 positive | 8 | 8
  Ki67 >=30%: number analyzed (Participants) | 71 | 65
  Ki67 >=30% | 21 | 13

6. Secondary Outcome: Number of Participants With Interval Breast Cancer
Description: Rate of interval breast cancer among those screened with tomosynthesis versus digital mammography as performed in a population based screening program.
Time Frame: 60 months from start up of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Breast Tomosynthesis | Digital Mammography
Number analyzed (Participants) | 14380 | 14369
Participants | 20 | 29

7. Other Pre Specified Outcome: Time Spent on Screen-Reading and Consensus Meetings
Description: The time spent on screen-reading and consensus will be compared for tomosynthesis versus digital mammography
Time Frame: 24 months from start up of the trial
Population: Interim analysis performed on study population from the first year of the trial (2016). All cases were screen-read by two radiologist, however not all were discussed at consensus.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Digital Breast Tomosynthesis | Digital Mammography
Number analyzed (Participants) | 7037 | 7052
seconds
  Initial screen reading | 70.5 (54.4) | 41.3 (49.6)
  Consensus reading: number analyzed (Participants) | 447 | 513
  Consensus reading | 192.1 (118.1) | 131.9 (79.2)

8. Other Pre Specified Outcome: Mammographic Features of Screen-Detected Breast Cancer
Description: as for outcome 5
Time Frame: 36 months from start up of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Breast Tomosynthesis | Digital Mammography
Number analyzed (Participants) | 95 | 87
Participants
  Spiculated mass | 35 | 16
  Indistinct mass | 16 | 16
  Calcifications | 13 | 20
  Architectural distortion | 10 | 7
  Asymmetry | 7 | 12
  Mass with calcifications | 7 | 11
  Circumscribed mass | 5 | 2
  Obscured mass | 1 | 3
  Associated features | 1 | 0

9. Other Pre Specified Outcome: Radiation Doses When Screening With Tomosynthesis Versus Digital Mammography
Description: Radiation doses will be measured for screening with tomosynthesis and digital mammography by an automated software, in milligray (mGy).
Time Frame: 24 months from start up of the trial
Population: Interim analysis performed on study population from the first year of the trial (2016). Not all women had available information on radiation dose.
Measure: Mean (Standard Deviation); unit: mGy
Arm/Group | Digital Breast Tomosynthesis | Digital Mammography
Number analyzed (Participants) | 6957 | 6972
mGy | 2.96 (0.62) | 2.95 (0.38)

ADVERSE EVENTS:
Time Frame: Participant were followed for two years after the recruitment period for the study ended (December 31st 2017) to collect data on adverse events. Reporting of adverse events are not yet complete as we rely on data from the Norwegian Cause of Death Registry.
Arm/Group | Digital Breast Tomosynthesis | Digital Mammography
All-Cause Mortality (participants affected / at risk) | 2/14734 | 2/14719
Serious Adverse Events (participants affected / at risk) | 0/14734 | 0/14719
Other Adverse Events (participants affected / at risk) | 0/14734 | 0/14719

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT02835625/Prot_SAP_001.pdf